CLINICAL TRIAL: NCT00000781
Title: A Randomized, Double-Blind, Four-Arm Study Comparing Combination Nucleoside, Alternating Nucleoside, and Triple-Drug Therapy for the Treatment of Advanced HIV Disease (CD4 <= 50/mm3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 193A; 11169 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; Nevirapine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Nevirapine; Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Nevirapine
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To determine the relative clinical efficacy of zidovudine ( AZT ) plus didanosine (ddI), AZT plus zalcitabine ( ddC ), AZT alternating monthly with ddI, and AZT/ddI plus nevirapine in HIV-infected patients with advanced disease.

The rapid emergence of resistant HIV strains has been observed in patients receiving monotherapy with a nucleoside analog or non-nucleoside reverse transcriptase inhibitor. Use of combination therapy with two nucleoside drugs or convergent combination therapy with two nucleosides and a non-nucleoside RT inhibitor may minimize the evolution of these resistant HIV strains. Since toxicity is a major problem in patients with advanced disease who are receiving combination nucleoside therapy, alternating the two drugs may provide a way of retaining several benefits of combination therapy while minimizing the increased toxicity.

DETAILED DESCRIPTION:
The rapid emergence of resistant HIV strains has been observed in patients receiving monotherapy with a nucleoside analog or non-nucleoside reverse transcriptase inhibitor. Use of combination therapy with two nucleoside drugs or convergent combination therapy with two nucleosides and a non-nucleoside RT inhibitor may minimize the evolution of these resistant HIV strains. Since toxicity is a major problem in patients with advanced disease who are receiving combination nucleoside therapy, alternating the two drugs may provide a way of retaining several benefits of combination therapy while minimizing the increased toxicity.

Patients are randomized to receive either AZT/ddC, AZT/ddI, AZT alternating monthly with ddI, or AZT/ddI/nevirapine. Patients are evaluated at week 0 and every 4 weeks thereafter for 2 years. Pharmacologic, virologic, and macroneurologic substudies will be conducted. Patients who are already enrolled on protocol ACTG 193 will be given the option of continuing on their originally assigned ACTG 193 therapy for an additional 6 months or undergoing re-randomization to one of the four treatment arms on ACTG 193A.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis.

Allowed:

* Erythropoietin maintenance.
* G-CSF and GM-CSF.
* Prophylaxis for Mycobacterium avium intracellulare.
* Antifungal prophylaxis or treatment with specific drugs.
* Maintenance therapy for opportunistic infection.
* Over-the-counter medications or alternative therapies such as vitamins and herbs.
* Antibiotics as clinically indicated.
* Steroids for < 21 days for acute problems.
* Antipyretics, analgesics, allergy medication, antidepressants, sleep medications, oral contraceptives, or other appropriate medications.

Concurrent Treatment:

Allowed:

* Radiation therapy for cutaneous Kaposi's sarcoma.
* Acupuncture.

Patients must have:

* Documented HIV infection.
* CD4 count <= 50 cells/mm3.
* Either no prior nucleoside therapy OR a history of prior nucleoside therapy in the absence of high-grade intolerance.
* Life expectancy of at least 6 months.
* Consent of parent or guardian if < 18 years of age.
* Normal chest x-ray at baseline or within 6 months prior to study entry in the absence of new pulmonary or cardiac symptoms (per 12/28/94 amendment).

NOTE:

* Patients who withdrew from protocol ACTG 193 therapy prior to activation of ACTG 193A are not eligible.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Abnormal baseline chest x-ray.
* New pulmonary or cardiac symptoms.
* Psychological or emotional problems sufficient to prevent compliance with study medication.

Concurrent Medication:

Excluded:

* Systemic chemotherapy for malignancy.
* Acute or induction therapy for opportunistic infection.
* Antiretroviral drugs other than study drugs.
* Biological response modifiers.
* Erythromycin, phenytoin, phenobarbital, warfarin, or coumadin.

Patients with the following prior conditions are excluded:

* History of recurrent grade 3 or greater toxicity to AZT, ddI, or ddC on two or more occasions.
* Evidence of active pulmonary disease within 6 months prior to study entry.
* History of grade 3 or worse peripheral neuropathy.
* History of acute or chronic pancreatitis.

Prior Medication:

Excluded:

* Prior nevirapine.

Excluded within 7 days prior to study entry:

* Acute therapy for opportunistic infection (maintenance therapy is permitted).
* Acute systemic therapy for a nonopportunistic infection or other medical condition.
* Antiretroviral drugs other than AZT, ddI, or ddC.
* Biological response modifiers.
* d4T therapy.
* Nucleosides other than those used in the study.
* Antibiotics containing clavulanate potassium.

Prior Treatment:

Excluded:

* More than 4 units of blood in a 30-day period.

Active alcohol or drug abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1292
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry WK, Study Chair; Kahn JO, Study Chair; Balfour HH, Study Chair
Locations (96):
- United States (95):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hosp of Los Angeles, Los Angeles, California
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Huntington Memorial Hosp / Children's Hosp of Los Angeles, Pasadena, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Olive View Med Ctr, Sylmar, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Denver Dept of Health and Hosps, Denver, Colorado
  - Mountain States Reg Hemo Ctr / Univ of Colorado, Denver, Colorado
  - Rose Med Ctr, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Yale Univ / New Haven, New Haven, Connecticut
  - HIV Ctr - District of Columbia Gen Hosp, Washington D.C., District of Columbia
  - Whitman - Walker Clinic / Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - George Washington Univ / Hershey Med Ctr, Washington D.C., District of Columbia
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of South Florida, Tampa, Florida
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Univ of Louisville / East Tennesee Comprehensive Hem Ctr, Louisville, Kentucky
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Worcester Memorial Hosp / Med Ctr of Cntrl MA-Memorial, Worcester, Massachusetts
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Dartmouth - Hitchcock Med Ctr / Med Ctr Cntrl Massachusetts, Lebanon, New Hampshire
  - Robert Wood Johnson Med School / Hershey Med Ctr, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Adirondack Med Ctr at Saranac Lake, Albany, New York
  - Albany Med College / Division of HIV Medicine A158, Albany, New York
  - Mid - Hudson Care Ctr, Albany, New York
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - North Shore Univ Hosp, Manhasset, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Clare's Hosp and Health Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr / Hemophilia Treatment Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Comprehensive Health Care Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Drug Treatment Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Family Health Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Samaritan Village Inc / Bronx Municipal Hosp, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Kentucky Lexington, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Columbus Children's Hosp, Columbus, Ohio
  - Med College of Ohio, Toledo, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Saint Michael's Med Ctr / Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Girard Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Med Univ of South Carolina / UNC, Charleston, South Carolina
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Meharry Med College, Nashville, Tennessee
  - Univ of Texas Galveston, Galveston, Texas
  - Univ Texas Health Science Ctr / Univ Texas Med School, Houston, Texas
  - Univ of Washington, Seattle, Washington
  - Northern Wisconsin Hemophilia Ctr / Saint Vincent's Hosp, Green Bay, Wisconsin
  - Great Lakes Hemophilia Foundation, Wauwatosa, Wisconsin
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Henry K, Erice A, Tierney C, Balfour HH Jr, Fischl MA, Kmack A, Liou SH, Kenton A, Hirsch MS, Phair J, Martinez A, Kahn JO. A randomized, controlled, double-blind study comparing the survival benefit of four different reverse transcriptase inhibitor therapies (three-drug, two-drug, and alternating drug) for the treatment of advanced AIDS. AIDS Clinical Trial Group 193A Study Team. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Dec 1;19(4):339-49. doi: 10.1097/00042560-199812010-00004. PMID 9833742
- [Background] Price RW, Yiannoutsos C, Zaborski L, Kmack A, Henry K, Tierney C, Clifford D. Neurological substudies of ACTG protocol 193A: quantitative neurological performance measures and treatment outcomes. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:176 (abstract no 516)
- [Background] Robinson P, Cotton D, Curry R, Henry K, Hall D, Myers M. Analysis of nevirapine (NVP) effect on clinical endpoints (CEs) of HIV progression or death in ACTG trial 193A. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:210 (abstract no 700)
- [Background] Henry K, Tierney C, Kahn J, Balfour H, Jiang Q, Kmack A, Fischl M. A randomized, double-blind, placebo-controlled study comparing combination nucleoside and triple therapy for the treatment of advanced HIV disease (CD4 less than or equal to 50/mm(3)). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:207 (abstract no LB6)
- [Background] Coplan P, Nikas A, Saah A, Nessly M, Doll L, Leavitt R, Benson J, Guess H. No association observed between indinavir therapy for HIV/AIDS and myocardial infarction in 4 clinical trials with 2,825 subjects. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:191 (abstract no 658)
- [Background] Erice A, Tierney C, Balfour HH Jr, Liou S, Kahn JO, Henry WK. Virologlc effect of therapy with reverse transcriptase inhibitors (RTIs) in patients with AIDS and less than 50 CD4+ T cells per mm(3): a substudy of ACTG 193a. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:204 (abstract no 662)
- [Background] Price RW, Yiannoutsos CT, Clifford DB, Zaborski L, Tselis A, Sidtis JJ, Cohen B, Hall CD, Erice A, Henry K. Neurological outcomes in late HIV infection: adverse impact of neurological impairment on survival and protective effect of antiviral therapy. AIDS Clinical Trial Group and Neurological AIDS Research Consortium study team. AIDS. 1999 Sep 10;13(13):1677-85. doi: 10.1097/00002030-199909100-00011. PMID 10509569